CLINICAL TRIAL: NCT06163963
Title: Sentinel Lymph Node Mapping with Double Tracer and Double Injection Sites in Early-Stage Endometrium Cancer
Brief Title: Sentinel Lymph Node in Early-Stage Endometrium Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/2015
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2023-12

CONDITIONS: Sentinel Lymph Node; Endometrial Cancer
Keywords: double tracer, endometrial cancer, sentinel lymph node
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: A single arm interventional study aiming at the comparison of the effectiveness of detection for sentinel lymph node biopsy using double tracer compared to classic single tracer in early stage endometrial cancer. So, we aimed to investigate whether the sentinel lymph node detection rates may be improved with double tracer injected at two different sites (charcoal carbon black dye injected in subserosa and ICG injected into cervix) compared to standard single tracer injected in early-stage endometrial cancer, especially the para-aortic sentinel lymph nodes. Sterile charcoal carbon black dye is an agent previously used for sentinel lymph node detection in various cancers such as breast cancer.
  Sentinel lymph node detection rates of each region (pelvic, obturator, inframesenteric para-aortic, supra-mesenteric - infrarenal para-aortic), bilaterality/ unilaterality and staining with single or double tracer will be discussed compared to literature data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sentinel Lymph Node Mapping With Double Tracer in Endometrium Cancer (Single Arm) (Experimental): Sentinel Lymph Node Mapping With Double Tracer and Double Injection Sites in Early-Stage Endometrium Cancer (Single Arm)
  Interventions: Diagnostic Test: Sentinel Lymph Node Mapping With Double Tracer and Double Injection Sites in Early-Stage Endometrium Cancer; Diagnostic Test: charcoal injection to uterus to map sentinel lymph nodes

INTERVENTIONS:
Diagnostic Test: Sentinel Lymph Node Mapping With Double Tracer and Double Injection Sites in Early-Stage Endometrium Cancer — This is a single arm interventional prospective study. Sentinel lymph node detection rate of the tracer injected in cervix (ICG- indocyanine green) before operation and the second tracer injected in uterine fundal subserosa (sterile charcoal black) at the start of operation are investigated. It is anticipated that additional tracer used in the uterine serosa may overcome the insufficiency (or increase the detection rate) of the standard single tracer injected in cervix for detection rate of sentinel lymph nodes, especially in paraaortic sentinel lymph nodes.
Diagnostic Test: charcoal injection to uterus to map sentinel lymph nodes — During surgery for endometrial cancer, charcoal injection to uterus to map sentinel lymph nodes in para aortic area besides the classic ınjection of indocyanine green for pelvic sentinel lymph node mapping.

SUMMARY:
The aim of this prospective study is to investigate whether the detection rate of sentinel lymph node (SLN) with double tracer injected at two different sites may be increased compared to the standard use of a single tracer with single site (cervix) injection in early-stage endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer. Although 85-90% of women are diagnosed at early stage, about 10-15% are diagnosed at advanced stages. Treatment and prognosis depends on the surgical staging of the apparently early stage disease including the evaluation of lymphatic status of the disease. Detection of positive lymph node upstages the apparently early stage endometrial cancer. However, systematic lymphadenectomy carries immediate and long term risks for patients including bleeding, massive transfusions, prolongation of operation time, serious major vessel and major abdominal organ injury and death. These risks are especially increased in para-aortic lymphadenectomy which is a part of staging procedure in apparently early stage endometrial cancer.

Sentinel lymph node biopsy (SLNB) procedure is the biopsy of one or two lymph node(s) which represents the lymph node basin draining the area of malignancy. This biopsy may potentially eliminate the need systemic pelvic / para-aortic lymphadenectomy which harbours potential complications. Although SLNB became an standard procedure in endometrial cancer, available data on the SLNB in endometrial cancer is variable. The relevant literature suggests that the detection rate of sentinel lymph node using various tracer agents are between %70-98, even with lower for bilateral pelvic detection and para-aortic sentinel lymph node(s). The most commonly used tracer agents are methylene blue, radiolabeled colloid technetium 99 (Tc99), isosulfan blue and fluorescent indocyanine green. Although subserosal, intramyometrial uterine injections and peritumoral injections using hysteroscopy with different tracers and different detection rates have been used, cervical injection with ICG is the most favoured and standard technique with highest pelvic SLN detection rates. However, the para-aortic SLN detection rates are not satisfactory with a single tracer injected into cervix which may be critical especially in high grade endometrioid, serous and clear cell histological types.

So, investigators aimed to investigate whether the sentinel lymph node detection rates may be improved with double tracer injected at two different sites (charcoal carbon black dye injected in subserosa and ICG injected into cervix) compared to standard single tracer injected in early-stage endometrial cancer, especially the para-aortic sentinel lymph nodes. Sterile charcoal carbon black dye is an agent previously used for sentinel lymph node detection in various cancers such as breast cancer.

Technically, 2 mL indocyanine green with sterile water is injected at 3 and 9 o'clocks (each 1 mL) of cervix before the start of laparoscopic operation. Additionally, 2-4 mL of sterile charcoal carbon black dye is carefully injected just beneath the serosal layer at uterine fundus bilaterally avoiding intravascular injection This is done classically during laparoscopy by a spinal needle introduced under optical supervision after all optical and operative instruments are entered. 10-15 minute interval is allowed before the start of harvesting sentinel lymph nodes in pelvic and paraaortic region.

ELIGIBILITY:
Inclusion Criteria:

1. Must have preoperative histologic diagnosis of endometrial carcinoma
2. Must be in early stage ( stage1 and 2) endometrial carcinoma radiologically and clinically
3. Must have written informed consent

Exclusion Criteria:

1. Possible allergic reaction to commonly used drugs
2. Medical or surgical contraindications for comphrensive staging
3. Preoperative or intraoperative findings of advanced endometrial cancer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female - endometrial carcinoma
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel lymph nodes with double tracer in early stage endometrial carcinoma | From the day of surgery to final pathology report (2 weeks)
  Detection rates of sentinel lymph nodes for both tracers in every pelvic and paraaortic lymph node basin are the primary outcome of the study.Sentinel lymph node detection rates of each region (pelvic, obturator, inframesenteric para-aortic, supra-mesenteric - infrarenal para-aortic), bilaterality/ unilaterality and staining with single or double tracer will be discussed compared to literature data.

CONTACTS AND LOCATIONS:
Overall Officials: Samet TOPUZ, PROF. DR., Study Director — ISTANBUL UNİVERSİTY MED FAC DEPT. OF OBSTET AND GYNECOL. DIVISION OF GYNECOLOGİC ONCOLOGY
Locations (1):
- Istanbul University Medical Faculty Dept. of Obstet Gynecol, Division of Gynecologic Oncology, Istanbul, Istanbul / Turkey, Turkey (Türkiye)

REFERENCES:
- [Background] Crosbie EJ, Kitson SJ, McAlpine JN, Mukhopadhyay A, Powell ME, Singh N. Endometrial cancer. Lancet. 2022 Apr 9;399(10333):1412-1428. doi: 10.1016/S0140-6736(22)00323-3. PMID 35397864
- [Background] Cibula D, Oonk MH, Abu-Rustum NR. Sentinel lymph node biopsy in the management of gynecologic cancer. Curr Opin Obstet Gynecol. 2015 Feb;27(1):66-72. doi: 10.1097/GCO.0000000000000133. PMID 25502426
- [Background] Lee YC, Lheureux S, Oza AM. Treatment strategies for endometrial cancer: current practice and perspective. Curr Opin Obstet Gynecol. 2017 Feb;29(1):47-58. doi: 10.1097/GCO.0000000000000338. PMID 27941361
- [Background] van den Heerik ASVM, Horeweg N, de Boer SM, Bosse T, Creutzberg CL. Adjuvant therapy for endometrial cancer in the era of molecular classification: radiotherapy, chemoradiation and novel targets for therapy. Int J Gynecol Cancer. 2021 Apr;31(4):594-604. doi: 10.1136/ijgc-2020-001822. Epub 2020 Oct 20. PMID 33082238
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221